CLINICAL TRIAL: NCT00195078
Title: Phase I-II Study of ZD1839 (IRESSA®), Cisplatin, and External-Beam Radiation Therapy in Patients With Locally Advanced, Non-Metastatic, Squamous Cell Carcinoma of the Head and Neck
Brief Title: Safety Trial of IRESSA, Cisplatin and Radiation Therapy for Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0404-218
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; squamous cell carcinoma of the oral cavity; squamous cell carcinoma of the oropharynx; squamous cell carcinoma of the larynx; squamous cell carcinoma of the hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: ZD1839 (IRESSA)
Drug: Cisplatin
Procedure: Radiation Therapy

SUMMARY:
The purpose of this study is to find out whether adding ZD1839 to standard treatment (Cisplatin and Radiation Therapy) of unresectable head and neck cancers is better than cisplatin and radiation alone.

DETAILED DESCRIPTION:
This is a Phase I-II, open-label, dose-escalation study in subjects with advanced head or neck cancer. Subjects will receive daily ZD1839 during a course of standard radiation therapy accompanied by cisplatin.

Subjects are adults with Stage III-IV squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx, who are in medically stable condition, with an Eastern Cooperative Oncology Group (ECOG) Performance Status of £ 1, stable hepatic and bone marrow function, and a life expectancy of at least 6 months. Subjects should have no previous cancer history (with the exception of squamous cell carcinoma of the skin or cervical cancer in situ) and no prior treatment with radiation, chemotherapy, or definitive surgical therapy. Subjects in the Phase II portion of the trial must have measurable disease as defined by RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx. For the Phase II portion of the study: measurable disease as based on RECIST criteria.
* Stage III or IV disease, M0.
* Life expectancy > 6 months.

Exclusion Criteria:

* Known severe hypersensitivity to ZD1839 or any of the excipients of this product.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years, with the exception of squamous cell carcinoma of the skin or cervical cancer in situ.
* Previous treatment with radiation, chemotherapy, or definitive surgical therapy.
* Distant metastatic disease.
* Documented evidence of HIV infection (because the interaction of ZD1839 with Highly Active Anti-Retroviral Therapy [HAART] is unknown).
* Substance abuse or psychiatric problems that would interfere with compliance.
* Pregnancy or breast-feeding (women of child-bearing potential).
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2004-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To explore whether the addition of ZD1839 to standard treatment of unresectable head and neck cancers (i.e., cisplatin and radiation therapy) improves the clinical complete response rate (as measured by RECIST criteria).

SECONDARY OUTCOMES:
To determine the time to disease progression, duration of response, and 2?year disease-free survival in subjects with unresectable tumors of the head and neck after combined therapy with ZD1839, cisplatin, and radiation.
To determine the toxicities, and recovery from toxicities, of combined therapy with ZD1839, cisplatin, and radiation therapy.
To determine dose-limiting toxicity as well as the recommended Phase II dose of ZD1839 given concurrently with cisplatin and radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Keresztes, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States